CLINICAL TRIAL: NCT06453967
Title: Impact of Blood Glucose Levels on in ICU Morbidity and Mortality in Patients With Acute Decompensated Heart Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, salma hamdy mahmoud haridi, Assistant lecturer, Assiut University
Other Study IDs: 2024-04-22-001
Record Dates: First submitted 2024-04-15; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
Keywords: glucose variability
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: blood glucose levels — measurement of blood glucose level at admission ,during ICU admission and at discharge for patients with acute decompensated heart failure

SUMMARY:
To evaluate the effect of blood glucose level at admission and glucose variability during ICU admission and their effect on in-hospital morbidity and mortality in patients admitted with acute decompensated heart failure

DETAILED DESCRIPTION:
Stress hyperglycemia is a physiological response of blood glucose levels to stressful events or severe diseases through enhanced inflammatory or neuro-hormonal activation , typically reflecting the severity of the corresponding disease.

Diabetes mellitus may lead to hyperglycemia. However, it can happen as a result of stress hormones in crucial situations as well as in illness states, and is referred to as "Stress Hyperglycemia". Other names for this syndrome include "New onset Hyperglycemia", "In hospital Hyperglycemia", "Admission Hyperglycemia", "New Hyperglycemia", and "reactive Hyperglycemia". The prevalence of admission hyperglycaemia ranges from 25 to 50% depending on the hyperglycaemia definition cut-off adopted. The American Heart Association and the Endocrine Society Clinical Guidelines defined stress hyperglycaemia as a random plasma glucose level above 140 mg/dL at any given time for both diabetic and nondiabetic hospitalized patients.Studies have shown that an elevated admission blood glucose level, in correlation with a specific condition, such as: myocardial infarction, stroke, heart failure or pneumonia is associated with a higher in-hospital mortality, increased length of hospital stay, and a higher rate of in-hospital complications.

Heart failure (HF) is a complex clinical syndrome that results from structural or functional impairment of ventricular filling or ejection. Also, HF is a progressive condition with intermittent acute decompensation leading to poor prognosis despite established guideline-directed therapy.Acute decompensated heart failure is a common reason for frequent hospital admission and has been associated with increased short-term mortality and poor long-term prognosis. Admission hyperglycaemia can be useful in identifying high-risk group of acute heart failure or in the risk stratification of acute heart failure In addition to age, obesity and diabetes have been identified as important risk factors for heart failure, Heart failure often manifests as the first cardiovascular event in people with type 2 diabetes.Several potential mechanisms contributing to the development of heart failure in diabetes include renin-angiotensin-aldosterone system (RAAS) activation, mitochondrial dysfunction, oxidative stress, inflammation, changes in intracellular calcium homeostasis, increased formation of advanced glycation end products, and myocardial energy substrate alterations including increased free fatty acid utilization, decreased glucose utilization, and increased oxygen consumption, resulting in decreased cardiac efficiency .

Dysregulation of hyperglycemia and glycemic variability are associated with an increased risk of mortality in critically ill patients .

It is also to be noted that individuals with HF and pre-diabetes have a higher risk of all-cause mortality and cardiac outcomes compared to those with normoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted with acute decompensated heart failure will be recruited in the study.

Exclusion Criteria:

* Patients on chronic steroid therapy Patients diagnosed with right sided heart failure due to chest disease Patients with malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed as acute decompensated heart failure and admitted to critical care unit will be recurited in this study either diabetic or not
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of glucose variability during ICU admission on in-hospital morbidity and mortality in patients admitted with acute decompensated heart failure ▪ | 1 year
  Glycaemic variability can be measured by Standard deviation of glucose, Coefficient of variation of glucose, Mean amplitude of glucose excursion ,glycemic lability index

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Obeid Allah, Phd, Study Director — Assiut University

REFERENCES:
- [Background] Zhou Y, Liu L, Huang H, Li N, He J, Yao H, Tang X, Chen X, Zhang S, Shi Q, Qu F, Wang S, Wang M, Shu C, Zeng Y, Tian H, Zhu Y, Su B, Li S; WECODe Study Group. 'Stress hyperglycemia ratio and in-hospital prognosis in non-surgical patients with heart failure and type 2 diabetes. Cardiovasc Diabetol. 2022 Dec 26;21(1):290. doi: 10.1186/s12933-022-01728-w. PMID 36572923
- [Background] Djupsjo C, Kuhl J, Andersson T, Lundback M, Holzmann MJ, Nystrom T. Admission glucose as a prognostic marker for all-cause mortality and cardiovascular disease. Cardiovasc Diabetol. 2022 Nov 26;21(1):258. doi: 10.1186/s12933-022-01699-y. PMID 36435766
- [Background] Paolisso P, Foa A, Bergamaschi L, Angeli F, Fabrizio M, Donati F, Toniolo S, Chiti C, Rinaldi A, Stefanizzi A, Armillotta M, Sansonetti A, Magnani I, Iannopollo G, Rucci P, Casella G, Galie N, Pizzi C. Impact of admission hyperglycemia on short and long-term prognosis in acute myocardial infarction: MINOCA versus MIOCA. Cardiovasc Diabetol. 2021 Sep 24;20(1):192. doi: 10.1186/s12933-021-01384-6. PMID 34560876
- [Background] Lee HY, Oh BH. Paradigm Shifts of Heart Failure Therapy: Do We Need Another Paradigm? Int J Heart Fail. 2020 Apr 6;2(3):145-156. doi: 10.36628/ijhf.2020.0010. eCollection 2020 Jul. PMID 36262366
- [Background] Kattel S, Kasai T, Matsumoto H, Yatsu S, Murata A, Kato T, Suda S, Hiki M, Takagi A, Daida H. Association between elevated blood glucose level on admission and long-term mortality in patients with acute decompensated heart failure. J Cardiol. 2017 Apr;69(4):619-624. doi: 10.1016/j.jjcc.2016.05.013. Epub 2016 Aug 21. PMID 27554050
- [Background] Cho JY, Kim KH, Lee SE, Cho HJ, Lee HY, Choi JO, Jeon ES, Kim MS, Kim JJ, Hwang KK, Chae SC, Baek SH, Kang SM, Choi DJ, Yoo BS, Ahn Y, Park HY, Cho MC, Oh BH. Admission Hyperglycemia as a Predictor of Mortality in Acute Heart Failure: Comparison between the Diabetics and Non-Diabetics. J Clin Med. 2020 Jan 6;9(1):149. doi: 10.3390/jcm9010149. PMID 31935874
- [Background] Ceriello A, Catrinoiu D, Chandramouli C, Cosentino F, Dombrowsky AC, Itzhak B, Lalic NM, Prattichizzo F, Schnell O, Seferovic PM, Valensi P, Standl E; D&CVD EASD Study Group. Heart failure in type 2 diabetes: current perspectives on screening, diagnosis and management. Cardiovasc Diabetol. 2021 Nov 6;20(1):218. doi: 10.1186/s12933-021-01408-1. PMID 34740359
- [Background] Pop-Busui R, Januzzi JL, Bruemmer D, Butalia S, Green JB, Horton WB, Knight C, Levi M, Rasouli N, Richardson CR. Heart Failure: An Underappreciated Complication of Diabetes. A Consensus Report of the American Diabetes Association. Diabetes Care. 2022 Jul 7;45(7):1670-1690. doi: 10.2337/dci22-0014. PMID 35796765